CLINICAL TRIAL: NCT02226289
Title: Phase II Study of Bevacizumab-containing Regimen in Patients With Metastatic Colorectal Cancer Who Failed to Cytotoxic Treatment
Brief Title: Bevacizumab-containing Regimen for Metastatic Colorectal Cancer Failed to Cytotoxic Treatment
Acronym: BATTLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Associate Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BATTLE
Record Dates: First submitted 2014-08-25; First posted 2014-08-27 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Neoplasm; Colorectal Cancer; Metastatic Neoplasm
Keywords: bevacizumab; refractory; colorectal cancer; metastatic
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Neoplasm Metastasis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bevacizumab-containing (Experimental): bevacizumab with the latest received cytotoxic regimen
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — bevacizumab with the latest received cytotoxic regimen
  Other Names: Avastin

SUMMARY:
Bevacizumab, a humanized monoclonal antibody against vascular endothelial growth factor (VEGF), combined with fluoropyrimidine-based chemotherapy is now the standard first and second-line treatment for metastatic colorectal cancer. The efficacy of bevacizumab with cytotoxic agents in the third-line treatment of patients with mCRC is still unknown.

DETAILED DESCRIPTION:
This is a single arm, phase II, open-labelled clinical trial to evaluate the safety and efficacy of bevacizumab combined with cytotoxic agents in the treatment of patients with mCRC progressing under all available cytotoxic chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained.
* Subjects must be able to understand and willing to sign a written informed consent.
* Subjects > 18 years of age
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2.
* Histological or cytological diagnosis of adenocarcinoma of the colon or rectum.
* Subjects have unresectable metastatic lesions.
* Subjects failed to respond to oxaliplatin, irinotecan and fluorouracil.
* Subjects have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria measured within 4 weeks prior to registration.
* Leukocytes ≥ 3.0 x109/ L, absolute neutrophil count (ANC) ≥ 1.5 x109/ L, platelet count ≥ 100 x109/ L, hemoglobin (Hb) ≥ 9g/ dL.
* Total bilirubin ≤1.5 x the upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5 x ULN.
* Amylase and lipase ≤ 1.5 x the ULN.
* Serum creatinine ≤ 1.5 x the ULN.
* Calculated creatinine clearance or 24 hour creatinine clearance ≥ 50 mL/ min.

Exclusion Criteria:

* Any previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to this study.
* Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization.
* Major surgical procedure, open biopsy, or significant traumatic injury within 4 weeks before start of study medication.
* Uncontrolled hypertension. (systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg despite optimal medical management).
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months before start of study medication.
* Any evidence of active infection.
* Known history of human immunodeficiency virus (HIV) infection.
* History of bleeding diathesis or coagulopathy.
* History of interstitial pneumonitis or pulmonary fibrosis
* Pregnancy or lactation at the time of study entry.
* Any history of or currently known brain metastases.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Any illness or medical conditions that are unstable or could jeopardize the safety of the subjects and his/her compliance in the study.
* Subjects with known allergy to the study drugs or to any of its excipients.
* Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | Baseline and 6 weeks
  Percentage of tumor regression

SECONDARY OUTCOMES:
Overall survival | From date of treatment until the date of death of any cause, assessed up to 48 months
  From date of treatment until the date of death of any cause
Progression free survival | From date of treatment until the date of disease progression, assessed up to 48 months
  From date of treatment until the date of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Ping Lan, Ph D, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No